CLINICAL TRIAL: NCT06983002
Title: Affect Consciousness (AC) as an Integrated add-on Component in Mentalization-based Group Treatment for Patients With Personality Disorder (PD)- a Mixed Method Explorative Study.
Brief Title: Bridging Affect Consciousness, Mentalization and Trauma- Exploring an Integrative Treatment Approach for Personality Disorder (PD).
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Helse Stavanger HF (Other Government)
Collaborators: Oslo University Hospital (Other); University of Oslo (Other); University College, London (Other); University of Stavanger (Other); Aalborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: RCT Personality Disorder STV25
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Personality Disorder, Borderline; Personality Trait; Personality Disorder; Personality Type; Personality Disorder, Avoidant; Affect Consciousness; Mentalization; Reflective Functioning; PTSD; PTSD - Post Traumatic Stress Disorder; PTSD and Trauma-related Symptoms
Keywords: Affect Integration; RCT; Affect Consciousness; MBT; AvPD; BPD; Trauma; Personality Disorder (PD); Personality functioning; Emotional dysfunction; Bodily Awareness; Art Therapy
MeSH Terms: conditions — Borderline Personality Disorder; Personality Disorders; Stress Disorders, Post-Traumatic; Combat Disorders; Wounds and Injuries

STUDY DESIGN:
Intervention Model Description: The raters and staticians are blinded. Clinicians not involved in the experimental intervention for research purposes will be used.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group: AC-group intervention as Add- on group to MBT group therapy (Experimental): The study's sample (N >300 in the period 2025-2035) is randomised into a two-group comparative design, 50% with AvPD and 50% with BPD will participate in an Affect Consciousness (AC) group as a supplement to MBT, experiment group.
  Interventions: Behavioral: Experimental group: AC-group therapy intervention.
- Control group 1: Body Awareness Group as Add on group to MBT group therapy (Active Comparator): 25% with AvPD and 25% with BPD will participate in an Body Awareness group as a supplement to MBT as a control group.
  Interventions: Behavioral: Control group 1: Body Awareness Group.
- Control group 2: Art Psychotherapy group as ADD- on to MBT group therapy (Active Comparator): 25% with AvPD and 25% with BPD will participate in an Art Psychotherapy group as a supplement to MBT as a control group.
  Interventions: Behavioral: Control group 2: Art Psychotherapy group.

INTERVENTIONS:
Behavioral: Experimental group: AC-group therapy intervention. — The aim is to increase Affect consciousness and Affect integration with 15 two hour group session interventions. Interview for 4 central affect categories to become familiar with the questions/techniques is used pre and post group. Group meeting 1 presents the AC affect theory, 13 affect categories and the group program related to each individual group meeting. Group meetings 2-14 lectures on the current affect category, bodily attentional signals and inner mood/mental content, exploration of impact, handling and the signal function of emotions and non-verbal body language and verbal descriptions related to the desire and ability to express oneself. Group meeting 15 is evaluation, clarification, repetition and closure of the group. "On arrival" focus on disturbances (internal and external) for each participant and performance of four body awareness exercises is used. Therapeutic writings and listening to a piece of music shared by the participants in rotation are methods i
  Arms: Experimental group: AC-group intervention as Add- on group to MBT group therapy
Behavioral: Control group 1: Body Awareness Group. — The aim is to connect with and become more confident about the body experiences, needs and feelings, to gain an increased understanding of oneself. The Group consists of 15 group sessions. Group meeting 1 Introduces Body Awareness Therapy, group structure and content and focus on experiences and expectations. The practice of slow, simple movements for the whole body in a standing position, introduction of The Autonomous Compass model, giving an opportunity to figure out where to place themselves in the compass in the moment, exercise stimulating the feet and a relaxation exercise. Group meetings 2-14 focuses on a topic as grounding, balance, breathe, play, posture due to habitual positions, body language and emotions, self-compassion and boundaries, explored through experience by using various physical exercises, sharing body experiences and psychoeducation. Session 15 contains summary, evaluation and repetition.Reflection on the previous session and sharing homework is included.
  Arms: Control group 1: Body Awareness Group as Add on group to MBT group therapy
Behavioral: Control group 2: Art Psychotherapy group. — The aim is to keep an open "non-directive" psychodynamic and analytical approach to explore, discover and feel ownership of creativity as a form of expression. The group consists of 15 group sessions, where session 1-4 is setting the framework by presenting art mediums to be used collectively, creating security, a sense of community and solidarity sharing common challenges. Each individual is free to choose the motive and form of expression, with a high level of sharing and learning. Creative experiences made together on the use of art materials to convey the inner world, become the starting point for further creative exploration on a individual level with their inner selves in a self-developing therapeutic process. Session 1: Introduction to projection and how to read oneself into an object by using figures and sandplay. Sessions 2 - 4: How one can transfer, animate, or create personal expressions using collage, acrylic painting and clay.Groups 5-15 allows freedom to choo
  Arms: Control group 2: Art Psychotherapy group as ADD- on to MBT group therapy

SUMMARY:
Study background: Specialized Group Outpatient Clinic within specialist mental health services, tailoring two year group treatment programmes for severe Avoidant PD (AvPD) and Borderline PD (BPD) with Affect Consciousness (AC) targeting specific areas of emotional dysfunction. Aims: Our main hypothesis, adding AC to Mentalization- based treatment (MBT) to expand the breadth and depth of therapeutically productive work on affect, will aim to examine health indicators, processes and mechanisms of change in depth. The study will extracts preliminary data after 5 years and 10 years to investigate clinical change, variation and outcome during MBT for PD employing AC as add on to MBT. The study has a randomized controlled trail design, with MBT with or without AC as add-on. The RCT is grounded on original literature on Affect Theory, as a framework for understanding patient functioning, and MBT, framing the therapy.Implications: AC methodology as add on can lead to more tailored treatment programmes, service planning, allocation of resources, guidelines, ACI certification and method development for PDs.

DETAILED DESCRIPTION:
Randomized Controlled Trial (RCT) design from an observational longitudinal dataset. The study is part of the National Network of Personality Psychiatry. Repeated measurements of dependent variables during treatment will uncover how treatment conditions and dependent variables develop. The study's sample (N >300 from 2025-2035) is randomised into a two-group comparative design, 50% with AvPD and 50% with BPD will participate in an AC group as a supplement to MBT. 50% from each PD type will represent two control groups. The National Network of Personality Psychiatry (the Network) is providing systematic routines and clinical systems for facilitating quality PD assessment and evaluation during treatment, for outcome measures see table.

Analyses will be performed using IBM SPSS Statistics, Version 27.0. Advanced statistical methods for longitudinal analyses will mainly include linear mixed methods, both within- and between patient levels of prediction, with dependent variables based on patient- reported outcome measures, predictors and moderators based on clinical reported information on treatment condition and structured clinician evaluation of diagnoses.

The statistical power to detect a small to moderate effect size of d = 0.35 was estimated by statistician based on an expected drop-out rate of 12% with the necessary sample size for each group determined to be N 132. The level of statistical significance was set to 0.05. Using an independent samples t-test (one-tailed), our study's estimated power to identify the effect is 0.883 (or 88.3%).

A higher anticipated drop-out rate of 30%, adjusts sample size to N 105. The estimated power slightly decreases to 0.81, still surpasses the commonly accepted threshold of 0.80, suggesting sufficient power to detect a small to moderate effect.

Our choice of a one-tailed t-test aligns with the directional hypothesis that the group receiving AC in conjunction with MBT will show more beneficial effects than the control group.

Alternatively, employing a two-tailed test with the original drop-out rate of 12% yields a power of 80.8% for detecting an effect size of d=0.35.

Data collection is including all patients included in the two group programmes for AvPD and BPD.

The study context is a Spezialized Group Outpatient Clinic within mental health services in Norway.The Group Outpatient Clinic is tailoring evidence-based, long-term MBT group programmes for severe BPD, first psychoeducational introduction group followed by dynamic MBT, both manualized to promote the ability to mentalize or to maintain mentalization.

Customized MBT will be offered for AvPD using a new norwegian MBT manual designed for AvPD. Individual MBT frequency will be accounted for in the publications.

Theoretical perspectives; Affect Consciousness (AC) is assumed to reflect the capacity to utilize one's emotional experiences for adaptive purposes and ensure appropriate regulation of self- and interpersonal relationship. Affect Integration (AI) is the operationalization of the emotional dysfunction described in the AC construct, assumed to protect against the development of psychopathology. Affect Consciousness Interview (ACI) is operationalized as the degree of consciousness, tolerance, nonverbal and conceptional expression of 11 distinct affects. The concept of mentalizing is defined as the implicit or explicit imaginative mental activity enabling us to recognise, visualize, perceive and interpret behaviour in terms of intentional mental states.

The experiment intervention ,AC Group, is a manual-based psychotherapy to enhance AC and integrate distinct affect categories.

Data will extracted after five years, presenting preliminary data in publication, but series of publication is planned for after datacollection is completed (2035). Repeated measurements of dependent variables during treatment will uncover how treatment conditions and dependent variables develop.

Blinded health staff generated the random allocation sequence by lottery (June 2024) for the period of 10 years to prevent selection bias. Clusters were enrolled based on group formation (20 patients with AvPD and 20 with BPD, yearly inclusion spring and autumn).

Outcome measures:

The participants undergo extensive examination at baseline, repeated every six months before termination (2- years programmes), including assessments, diagnostics, interviews and self-report questionnaires. Treatment duration and adherence will be specified. All patients are diagnosed with SCID-5-PD and the Mini International Neuropsychiatric Interview (M.I.N.I.), confirmed by specialists in psychiatry/clinical psychology. PTSD will be assessed by use of a structured clinical interview (MINI) based on screening indicating PTSD.

Methodological considerations: A Risk and contingency plan will account for drop-outs, characteristics and reasons, and how this may have affected the results. A consort diagram will show the flow of participants, analyzed according to the "intention to treat" principle, including all participants, regardless of whether they completed the study, reducing attrition bias. Due to an estimated greater risk of drop-out for PD, we will report carefully. The study has stipulated N >300, estimated from national and international drop-out rates. Following patients over long-time spans can give unbalanced outcome due to incomplete participant evaluations. The statistical method is enabling high utilization of available longitudinal data. The randomisation on a cluster level is chosen due to ethical and social considerations, mixing vulnerable patients across groups. We are recruiting from one geographical area, where our clinic is the only clinic nationally systematically employing AC with MBT for research purposes, giving us no possibility to compare datasets from other units. "The Network" provides a large comparison group with standard MBT after RCT completion.

Satisfactory power analysis is estimated. Well-established assessments and interviews used give considerable strengths. Blinded health staff perform the randomization. All clinicians in the treatment will participate in a reliability test to ensure their fidelity to the MBT model, based on adherence and quality at the Quality Laboratory for Psychotherapy (the Lab), at Oslo University Hospital (OUS). The team of clinicians receives MBT-supervision weekly, representing a quality system. The "Network" is enabling a strong test battery and safe data storage in a quality registry, DN 2000. A total of 5 measurements provides strengths. To avoid reporting bias, CONSORT guidelines for pre-reporting RCT studies are followed, where ongoing monitoring can correct deviations. Reporting both significant and non-significant results will improve credibility and reliability and counteract publication bias. Extern providers are working on blinded datasets, Comorbidity will be accounted for and optional data give access to data missing in the "Network", ( for information on test battery see below).

Validated patient self-report measures are choosen.

1. . Affect Integration: Affect Consciousness Interview (ACI). Affect Integration Inventory (extended version) (AII). Difficulties in Emotion Regulation Scale (DERS) Toronto Alexithymia Scale (TAS-20), Brief Mentalized Affectivity Scale (B-MAS).
2. . Personality functioning: Level of Personality Scale- Brief form (LPFS-BF) Severity Indices of Personality Problems-118 (SIPP118) The Experiences in Close Relationship Scale (ECR).
3. .Reflective functioning: The Reflective Functioning Questionnaire (RFQ-54).
4. .Trauma: The Adult Attachment Interview (AAI) Post Traumatic Stress Disorder Check List 5 (PTSD CL5) International Trauma Questionnaire (ITQ) Questionnaire for the assessment of body experience (SKO). Childhood Trauma Questionaire (CTQ)
5. . Symptoms & Functioning: General Anxiety Disorder -7 (GAD-7) Patient Health Questionnaire -9 (PHQ9).

The RCT- study is part of The Norwegian Network for Personality Disorders (The Network), a quality register within Norwegian PD research providing systematic routines and clinical systems for facilitating better quality PD assessment and evaluation during treatment. "The Network" is a well-etablished cross-regional quality and research collaboration where currently 20 PD treatment units within specialist mental health services across Norway contribute. The quality register of aggregated multicenter data, also represent a security system generating individual clinical profiles for local patient evaluation and safe storage.

Group programmes: In MBT, the aim is to promote the ability to mentalize or to maintain mentalization. Evidence-based, long-term MBT treatment programme for severe BPD contain regular psychoeducational MBT introduction group followed by dynamic MBT. Severe and more complex conditions are recommended to work in a long-term framework. Customized MBT was offered for AvPD using a MBT manual designed for AvPD. Individual MBT was provided for the period of two years, where the frequency is accounted for in the flow chart presenting results.

The clinicians will participate in a treatment reliability test. The clinicians also participate in Mentalization- based video-supervision. The battery used from the "Network" DN2000 included both patient and clinician reports. Separate items on sociodemographic data will be part of the study.

Additional questionaires and interviews relevant for this study (ACI, AII, B-MAS and RFQ54) not included in DN2000 (Pedersen et al, 2022) was approved by the Regional Committee for Medical Research Ethics in the Western Norway.

1. outcome Emotional functioning:

   Study Objective: To evaluate changes in emotional functioning over a two-year period among patients with AvPD and BPD undergoing a manualized mentalization-based group therapy programme (MBT-G) with Affect Consciousness (AC) group intervention as add on. The study aims to assess the efficacy of AC in improving affect integration, alexithymia, and affective mentalization integrating self-report and interview-based instruments.

   Research Questions: 1. "What are the changes in emotional dysfunction after two-year MBT-G applying AC as a supplement?" 2. Are changes in affect integration, alexithymia, and mentalized affectivity associated with the duration of therapy? 3. Do patients with AvPD and BPD show differential patterns of emotional change across the intervention period?

   Hypotheses: 1. Hypothesis: We assume that AC, providing specific questions used flexibly as a framework for emotional exploration, works better in the clinic than MBT's biological model alone. Patients assigned to the AC group as add on to MBT-G will have profiles with increased emotional functioning, especially for AvPD. 2. Hypothesis: Improvements in emotional functioning will occur progressively over time. Variation in longitudinal course and treatment processes will correlate more strongly with overall severity than PD type. 3. Hypothesis: The pattern and magnitude of emotional change may differ by diagnostic group, where the decrease of affect integration affects the ability to mentalize to a greater extent for AvPD.

   Outcome measures: Emotional dysfunction will be assessed using five validated self- report instruments: the Affect Consciousness Interview (ACI), the Affect Integration Inventory (AII), the Toronto Alexithymia Scale (TAS-20), the Brief Mentalized Affectivity Scale (B- MAS), and the Difficulties in Emotion Regulation Scale (DERS). Together, these instruments provide a multi-dimensional and clinically meaningful assessment of emotional dysfunction, which is a core feature of PD and a key target of MBT-G. The instruments capture complementary but distinct dimensions of emotional functioning, conducted at five time points: baseline (T1), and at 6, 12, 18, and 24 months (T2-T5). To account for changes over time within-subject correlations and time-varying effects in emotional functioning mixed- effects models will be used.
2. outcome Personality functioning

   Study Objective: To investigate changes in personality functioning among patients diagnosed with AvPD and BPD undergoing a two-year mentalization-based group therapy program (MBT-G) with AC as add on. Personality functioning will be assessed using dimensional measures consistent with contemporary models of personality pathology.

   Research Questions: 1. Does participation in an AC group as add on to MBT-G lead to improvements in personality functioning as measured dimensionally over the two-year treatment period? 2. Are changes in personality functioning associated with changes in emotional functioning across time? 3. Do patients with AvPD and BPD show different trajectories in the development of personality functioning?

   Hypotheses 1. Hypothesis: Patients in the AC group will demonstrate higher improvement in personality functioning over time, 2. Hypothesis: Changes in personality functioning will be correlated with improvements in emotional functioning, suggesting shared therapeutic mechanisms of change. 3. Hypothesis: Differential patterns of change may emerge between diagnostic groups, with BPD patients showing greater improvement in self-identity and affect regulation, and AvPD patients showing greater changes in relational functioning.

   Outcome Measures: Personality functioning will be assessed using three validated dimensional instruments reflecting the Alternative Model for Personality Disorders (AMPD): Level of Personality Functioning Scale - Brief Form 2.0 (LPFS-BF 2.0), Severity Indices of Personality Problems - 118 (SIPP-118) and Experiences in Close Relationships Scale (ECR). Together, these instruments provide a comprehensive, dimensional, and theoretically grounded assessment of personality functioning. Assessments will be administered at five time points: baseline (T1), and at 6, 12, 18, and 24 months (T2-T5). Data will be analyzed using longitudinal mixed-effects models to account for within-subject correlations and time-varying effects.
3. outcome Reflective functioning

   Study Objective: To examine changes in reflective functioning-conceptualized as the capacity for mentalization-across a two-year of MBT-G for patients with AvPD and BPD.

   Research Questions 1. Does participation in AC group supplementary to MBT-G lead to changes in RF over the course of two years? 2. Are improvements in RF associated with changes in emotional functioning and personality functioning? 3. Do the diagnostic subgroups AvPD vs. BPD differ in their trajectories of change in RF during MBT-G?

   Hypotheses 1. Hypothesis: All patients will show an increase in RF indicated by movement toward optimal scores on the RFQ-54, from baseline to 24 months, but patients from the AC group will have higher increase in RF. 2. Hypothesis: Increases in RF will be positively correlated with improvements in emotional and personality functioning over time. 3. Hypothesis: Patients with AvPD will show a steeper increase in RF compared to those with BPD, due to higher initial dysregulation and the targeted focus of MBT on affective mentalization.

   Outcome Measure: Reflective functioning will be assessed using the Reflective Functioning Questionnaire (RFQ-54), Scores will be analyzed longitudinally across five time points, baseline (T1), and at 6, 12, 18, and 24 months (T2-T5) using mixed-effects modeling to account for changes over time and potential interaction effects with diagnoses and other outcome variables. The RFQ-54's dimensional nature supports fine-grained analyses of individual trajectories of Mentalization-related change.
4. outcome Trauma

   Study Objective: To investigate the role of traumatic experiences-developmental, relational, and event-related-in shaping psychological functioning in patients with AvPD and BPD, and to examine how trauma-related symptoms and bodily experiences develop over the course of a two-year MBT-G intervention.

   Research Questions: 1. How do patterns of attachment and trauma symptomatology interact at baseline? 2. Do symptoms of post-traumatic stress and disturbances in self-organization (DSO) decrease over the course of MBT-G? 3. Are changes in trauma-related symptoms associated with changes in reflective functioning, emotional regulation, or personality functioning?

   Hypotheses: 1. Hypothesis: Patients will have a reduction in trauma-related symptoms-measured by PCL-5, ITQ and SKO from baseline to 24 months. 2. Hypothesis: Changes in trauma symptoms over time will correlate with improvements in emotional functioning and reflective functioning, suggesting overlapping treatment mechanisms. 3. Hypothesis: BPD participants will report higher levels of childhood trauma, unresolved attachment, and PTSD symptoms than AVPD participants at baseline.

   Outcome Measures: Traumatic exposure and symptomatology will be measured using a multimethod approach, integrating self-report and interview-based instruments. Five instruments capturing various aspects of traumatic experience and symptomatology: The Adult Attachment Interview (AAI), Post Traumatic Stress Disorder Check List 5 (PTSD CL 5), International Trauma Questionnaire (ITQ), Childhood Trauma Questionaire (CTQ) and Questionnaire of body experience (SKO) conducted at baseline (T1) and at 6-month intervals (T2-T5). Statistical analyses will include longitudinal modeling to assess changes over time and mediation/moderation analyses to explore relationships between trauma, emotional functioning, and personality outcomes.
5. outcome Symptoms & Functioning

Study Objective: To investigate the severity and course of anxiety and depressive symptoms in patients with AvPD and BPD participating in a two-year MBT-G.

Research Questions: 1. Do symptoms of anxiety and depression decrease over time during participation in MBT-G? 2. Are reductions in symptom severity associated with improvements in emotional functioning, personality functioning, or reflective functioning? 3. Do individuals with AVPD and BPD differ in their symptom profiles or treatment trajectories?

Hypotheses: 1. Hypothesis: Patients will show reductions in self-reported anxiety (GAD-7) and depressive symptoms (PHQ-9) from baseline to 24 months. 2. Hypothesis: Symptom reductions will be positively associated with improvements in emotional regulation, reflective functioning, and personality functioning. 3. Hypothesis: BPD participants will report higher baseline symptom severity and show greater fluctuations over time, while AVPD participants will report more stable but persistent symptom patterns.

Outcome Measures: Symptom severity and general psychological functioning will be assessed using the Generalized Anxiety Disorder-7 (GAD-7) and the Patient Health Questionnaire-9 (PHQ-9), validated self-report instruments. Baseline assessment will provide symptom profiles across the AVPD and BPD groups, helping to characterize the clinical burden in each diagnostic subgroup. Treatment response will be tracked over five time points (baseline, 6, 12, 18, and 24 months). Sustained reductions in GAD-7 and PHQ-9 scores will be interpreted and correlations with other outcome domains will be explored to examine interrelations between symptom relief and core personality processes. Changes over time will be analyzed using mixed-effects models to account for within-subject correlations and time-varying effects.

ELIGIBILITY:
Inclusion Criteria: Participation in a MBT programme for severe AvPD and/or BPD 2025-2035. Half the participants join an AC group as add on to standard MBT based on randomisation on a cluster level, 25 % of the rest of the 50% representing the control group patientsample join an Body Awareness Group as add on to proper MBT and the last 25%, representering the control group participates in an Art psychotherapy group as add on to MBT, Norwegian language proficiency, age 20- 40 years.

Exclusion Criteria: Diagnosed with schizotypal or antisocial PD, psychotic- or bipolar I disorder, pervasive developmental disorder, ongoing drug/ alcohol dependence, organically contingent symptoms and/or attention deficit hyperactivity disorder if not effectively treated with medication.

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-05-19 (Estimated); Primary Completion 2029-05-19 (Estimated); Study Completion 2035-04-19 (Estimated)

PRIMARY OUTCOMES:
Changes in emotional dysfunction, ACI evaluation | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  The Affect Consciousness Interview (ACI), scale 1-9. Higher scores indicate more integrated and conscious affective functioning, whereas lower scores suggest difficulties in affect regulation or alexithymic traits.
Changes in emotional dysfunction, All self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Affect Integration Inventory (AII), rating 112 items on a 10-point Likert scale (0 = does not fit at all, 9 = fits perfectly), where lower scores indicate lower affect integration across specific emotions.
Changes in emotional dysfunction, TAS-20 self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Toronto Alexithymia Scale (TAS-20), rating 20 items on a 5-point Likert scale (1 = strongly disagree, 7 = strongly agree), where total scores: ≥61 = high alexithymia, 52-60 = possible alexithymia, ≤51 = non-alexithymic
Changes in emotional dysfunction, B-MAS self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Brief Mentalized Affectivity Scale (B-MAS), rating 12 items on a 5-point Likert scale (1 = strongly disagree, 7 = strongly agree), where lower scores reflect suggest difficulties in affective self- reflection and regulation.
Changes in emotional dysfunction, DERS self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Difficulties in Emotion Regulation Scale (DERS), rating 36 items on a 5-point Likert scale (1 = almost never, 7 = almost always), where higher scores reflect higher level of problems with regulating emotions.
Changes in personality functioning, LPFS-BF self-report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Level of Personality Functioning Scale - Brief Form 2.0 (LPFS-BF 2.0), rating 12 items on a 4-point Likert scale (0 = not at all true, 3 = completely true), where higher scores indicates higher levels of personality dysfunction.
Changes in personality functioning, SIPP-118 self-report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Severity Indices of Personality Problems - 118 (SIPP-118), ratring 118 items in a 4-point Likert scale (1 = fully disagree, 4 = fully agree), where higher scores reflect better adaptive personality functioning.
Changes in personality functioning, ECR self-report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Experiences in Close Relationships Scale (ECR), rating 36 items on a 7-point Likert scale (1 = strongly disagree, 7 = strongly agree), where higher scores indicate higher levels of attachment-related anxiety and attachment-related avoidance.
Changes in reflective functioning, RFQ-54 self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Reflective Functioning Questionnaire (RFQ-54), rating 54 items on a 7-point Likert scale (1 = completely disagree to 7 = completely agree), where higher scores indicate reduced reflective functioning.
Role of attachment related trauma - AAI | At time of inclusion (baseline), and at 6, 12 18 and 24 months
  The Adult Attachment Interview (AAI) uses the AAI Scoring System related to: coherence of mind (scale 1-9), unresolved loss (scale 1-9), unresolved trauma (scale 1-9), idealization of parents (scale 1-9), anger and passivity (scale 1-9), derogation, fear, and lack of memory (scale 1-9), and classifies the individual into categories of: autonomous/secure, dismissing, preoccupied, or unresolved/disorganized. This is to determine the individual's state of mind regarding early attachment experiences and related trauma symptoms.
Changes in PTSD symptoms, PCL-5 self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Post-Traumatic Stress Disorder Checklist for DSM-5 (PCL-5), rating 20 items 5-point Likert scale (0 = not at all, 4 = extremely), , where higher scores indicate higher levels of PTSD symptoms and a score ≥31 suggests probable PTSD diagnosis.
Changes in PTSD and C-PTSD symptoms, ITQ self report | At time of inclusion (baseline) and at 24 months
  Self-report questionnaire: International Trauma Questionnaire (ITQ), rating 18 items on a 5-point Likert scale (0 = not at all, 4 = extremely), evaluating symptoms of Post Traumatic Stress Disorder (PTSD) and Complex PTSD (CPTSD) and whether the individual have these diagnoses.
Traumatic childhood experience, CTQ self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Childhood Trauma Questionnaire - Short Form (CTQ-SF), rating 28 items on a 5-point Likert scale (1 = never true, 5 = very often true), determining levels of early childhood maltreatment of emotional abuse, physical abuse, sexual abuse, emotional neglect and pysical neglect. Higher scores indicate greater exposure to developmental trauma.
Changes in subjective bodily experience and body image, SKO self report | At time of inclusion (baseline), and at 6, 12, 18, and 24 months
  Self-report questionnaire: Questionnaire of Body Experience (SKO), rating 64 items on a 6-point Likert scale (1 = never, 6 = All the time), where higher scores in negative dimensions indicates higher levels of dissociation, body alienation and/or trauma-related disturbances.
Changes in levels of anxiety, GAD-7 self report | At time of inclusion (baseline) and at 24 months
  Self-report questionnaire: Generalized Anxiety Disorder-7 (GAD-7), rating 7 items on a 4-point Likert scale (0 = not at all, 3 = nearly every day), where higher scores indicate higer levels of anxiety. A decrease of ≥4 points is considered a clinically significant improvement.
Changes in depression symptoms, PHQ-9 self report | At time of inclusion (baseline) and at 24 months
  Self-report questionnaire: Patient Health Questionnaire-9 (PHQ-9), rating 9 items on a 4-point Likert scale (0-3), where higher scores indicates higher levels of depression symptoms. A reduction of ≥5 points is considered clinically significant.

CONTACTS AND LOCATIONS:
Overall Officials: Ole Andrè Solbakken, Scientific Director/prof/PhD, Study Director — Section of Clinical Psychology at the Department of Psychology (PSI), Institute of Affect Theory and Psychotherapy group (IATP)The University of Oslo (UIO). Norway..; Inge Joa, PI/Associate professor/PhD, Principal Investigator — The Regional Network for Clinical Psychosis Research (Psyk Nett Vest), the Western Norway Regional Health Authority, Stavanger University Hospital (SUS).
Locations (1):
- Stavanger University Hospital, Stavanger, Rogaland, Norway

IPD SHARING:
Plan to Share IPD: Yes
The data associated with the Network for Personality Disorders (referred to as routine data with a separate Regional Ethical Committee (REC) approval through Network for Personality Disorders and Oslo University Hospital) will after end og study become a part of the network's anonymized database. The patients approve that routine data is converted to the Network's quality register upon written study consent.
  All other data, i.e. quantitative and qualitative additional data will be deleted after 10 years.